CLINICAL TRIAL: NCT05422001
Title: Low-dose KETamine as an Adjunct to MOrphine for Acute Pain in the ED: a Randomized, Double-blinded Clinical Trial
Brief Title: Low-dose KETamine as an Adjunct to MOrphine for Acute Pain in the ED
Acronym: KetMo
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Not able to recruit opioid tolerant patients as expected
Sponsor: University of Aarhus (Other)
Collaborators: Central Denmark Region (Other); Aarhus University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KetMO
Record Dates: First submitted 2022-05-27; First posted 2022-06-16 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Acute Pain; Opioid Use
Keywords: Low dose ketamine; Opioid use; Acute pain; Emergency Department
MeSH Terms: conditions — Acute Pain; Emergencies | interventions — Ketamine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention, low-dose ketamine (Experimental): Two 1 ml syringes with Esketamine (5 mg/ml) will be prepared and study drug will be administered as intravenous bolus dose, 0,1 mg/kg. The study drug will be administered after an intravenous morphine dose.
  Interventions: Drug: low dose ketamine
- Placebo (Placebo Comparator): Two 1 ml syringes with saline will be prepared and study drug will be administered as intravenous dose, same volume as if Esketamine. The placebo drug will be administered after an intravenous morphine dose.
  Interventions: Drug: Placebo (saline)

INTERVENTIONS:
Drug: low dose ketamine — Low dose ketamine 0.1 mg/kg Product: Esketamin "Orifarm" 5 mg/ml
  Arms: Intervention, low-dose ketamine
Drug: Placebo (saline) — Isotonic Saline
  Arms: Placebo

SUMMARY:
The KetMo study is an investigator-initiated, randomized, parallel group, double blinded trial investigating if ketamine as an adjunct to morphine improves pain treatment in the ED.

Patients in pain (assessed on NRS, 5 or more) will be randomized to low-dose ketamine or placebo as an adjunct to morphine. Patients with or without prior use of opioids will be randomized separately.

The primary outcome will be pain reduction, assessed on NRS, after 10 minutes. Secondary outcomes include pain reduction until 120 minutes after injection of study medicine, need for rescue opioid, side effects and patient- and provider satisfaction.

ELIGIBILITY:
Inclusion Criteria:

1. Emergency Department admission
2. Age ≥ 18 years
3. NRS ≥ 5
4. Stable vital signs defined as systolic blood pressure ≥ 90 mmHg, heart rate between 60 and 150 per minute, respiratory rate between 8 and 26 per minute, oxygen saturation greater than or equal to 92%

Exclusion Criteria:

1. Initial management by trauma-team
2. Systolic blood pressure ≥ 180mmHg, severe untreated arrhythmia, unstable angina, recent myocardial infarction (< 30 days), severe heart-failure (Ejection fraction < 40 %)
3. Symptoms of untreated hyperthyroidism
4. Cirrhosis with ascites
5. Known/suspected pregnancy or breastfeeding
6. Patients for whom consent is not obtainable or psychiatric forced treatment.
7. Previously enrolled in the trial
8. Psychiatric illness prior to admission defined as prior psychosis/schizophrenia
9. Untreated diagnosed glaucoma
10. Known hypersensitivity to ketamine or to any excipient or prior use of ketamine with a negative experience (i.e. hallucinations)
11. Patient clearly influenced by drugs or alcohol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2022-05-31 (Actual); Primary Completion 2023-08-15 (Actual); Study Completion 2023-08-15 (Actual)

PRIMARY OUTCOMES:
Pain reduction after 10 minutes assessed on numeric rating scale, NRS | 10 minutes
  Numeric Rating Scale, 0-10

SECONDARY OUTCOMES:
Pain intensity assessed on numeric rating scale, NRS | 120 minutes
Need for rescue opioid | 120 minutes
  any kind of opioid
Side effects | 120 minutes
  At each time point (10 min, 20 min, 30 min, 45 min, 60 min and 120) vital parameters are measured (Blood pressure, Respiratory Frequency, Saturation, Heart Rate) and the patient are asked if they experience nausea/vomiting, a dream like state/dissociation/out of body experience, anxiety or dizziness.
  Besides a objective RASS score +4 to -5 (combative/very agitated/agitated/restless/aler and calm/drowsy/light sedation/moderate sedation/deep sedation/unarousable
Patient satisfaction | 120 minutes
  Lickert scale
Provider satisfaction | 120 minutes
  Lickert scale
Comparison af pain reduction ( prior use of opioid vs no prior use of opioid | 120 minutes
Patient Rated Pain Relief | Patient are asked at timepoint 10 and timepoint 120
  6 point lickert scale - worse pain, no pain relief, little pain relief, moderate pain relief, good pain relief, complete pain relief.

CONTACTS AND LOCATIONS:
Overall Officials: Stine F Galili, MD, Principal Investigator — Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Aarhus N, Vælg En Region, Stat Eller Provins., Denmark

IPD SHARING:
Plan to Share IPD: Yes
Six month after the publication of the last results, all de-identified individual patient data will be made available for data sharing
Supporting Information: Study Protocol, SAP, Analytic Code

REFERENCES:
- See also: Related Info — https://recem.au.dk/ketmo

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan: Latest amendment (2023-05-26): https://cdn.clinicaltrials.gov/large-docs/01/NCT05422001/Prot_SAP_001.pdf
  • Statistical Analysis Plan: Updated statistical analysis plan before unblinding (2023-09-15): https://cdn.clinicaltrials.gov/large-docs/01/NCT05422001/SAP_002.pdf